CLINICAL TRIAL: NCT06547099
Title: Blood Amyloid, Tau, and Neurodegeneration Biomarkers and Prediction of Clinical Onset, Cognitive Decline, and Dementia Diagnosis
Brief Title: Study to Understand Novel Biomarkers in Researching Dementia
Acronym: SUNBIRD
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 202405156; R01AG061900 (NIH)
Record Dates: First submitted 2024-08-01; First posted 2024-08-09 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment; Dementia
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, buffy coat, red blood cells
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cognitively normal: Participants without symptoms of cognitive impairment will be followed up annually for potential cognitive changes, and will complete additional blood collections every two years.
  Interventions: Other: Research blood collection; Other: Cognitive assessments
- Cognitively impaired: For participants with symptoms of cognitive impairment, their medical providers will review the results of the research cognitive assessments and determine whether further testing (a clinical tau PET scan and choice of an amyloid PET, cerebrospinal fluid, or blood clinical test for amyloid plaques) is needed. Symptomatic participants will be followed up annually for research blood collections and cognitive assessments.
  Interventions: Diagnostic Test: Clinical tau PET; Diagnostic Test: Clinical amyloid test; Other: Research blood collection; Other: Cognitive assessments

INTERVENTIONS:
Diagnostic Test: Clinical tau PET — Tau PET (flortaucipir)
  Groups: Cognitively impaired
Diagnostic Test: Clinical amyloid test — Amyloid PET (florbetapir), CSF amyloid test, or blood amyloid test
  Groups: Cognitively impaired
Other: Research blood collection — Research blood assays for amyloid, tau, and neurodegeneration
Other: Cognitive assessments — Clinical Dementia Rating (CDR) or electronic Clinical Dementia Rating (eCDR); Montreal Cognitive Assessment (MoCA)

SUMMARY:
The purpose of this study is to determine the relationships between amyloid, tau, and neurodegeneration biomarkers in the blood and the presence of Alzheimer's disease (AD) pathology, clinical cognitive decline, and diagnosis. We aim to understand how well blood-based biomarkers can diagnose and predict Alzheimer's disease, which will help to further develop and validate blood tests for the disease.

DETAILED DESCRIPTION:
All participants who are eligible and provide informed consent will complete an initial study visit, which includes a research blood collection and cognitive assessments. Depending on the results of the cognitive assessments, participants will complete follow-up visits annually or biennially for additional cognitive testing, research blood collections, and potential clinical testing for Alzheimer's disease as determined by the participant's medical provider.

ELIGIBILITY:
Inclusion Criteria:

* At least 60 years of age
* 80% of the newly enrolled clinic-based cohort will have symptoms of forgetfulness, mild cognitive impairment, mild dementia, or Alzheimer's disease as determined by their medical chart and/or provider
* All SEABIRD participants will be invited to participate regardless of their cognitive status

Exclusion Criteria:

* Unable to perform one or more basic activities of daily living (eating, bathing, dressing, ambulating, toileting) due to cognitive impairment
* Uncontrolled hepatitis B, hepatitis C, or HIV at time of blood collection
* Taking a disease-modifying drug for AD at time of enrollment
* Blood transfusion in the last three months
* Unwilling or unable to participate in all study activities

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All participants who completed our prior study, the Study to Evaluate Amyloid in Blood and Imaging Related to Dementia (SEABIRD, NCT03899844), will be invited to join SUNBIRD. We will also recruit approximately 1000 new participants from Washington University and Barnes-Jewish Hospital affiliated clinics in the greater St. Louis metropolitan area.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Area under the curve (AUC) of plasma amyloid-beta 42/40 in predicting amyloid PET status | Baseline
Area under the curve (AUC) of plasma %p-tau217 in predicting amyloid PET status | Baseline
Area under the curve (AUC) of plasma p-tau217 in predicting tau PET status | Baseline
Area under the curve (AUC) of plasma p-tau205 in predicting tau PET status | Baseline
Area under the curve (AUC) of plasma neurofilament light in predicting tau PET status | Baseline
Area under the curve (AUC) of plasma %p-tau205 in predicting clinical diagnosis | Baseline, 1 year, 2 years, 3 years, 4 years, 5 years
Area under the curve (AUC) of plasma %p-tau217 in predicting clinical diagnosis | Baseline, 1 year, 2 years, 3 years, 4 years, 5 years
Area under the curve (AUC) of plasma amyloid-beta 42/40 in predicting clinical diagnosis | Baseline, 1 year, 2 years, 3 years, 4 years, 5 years
Area under the curve (AUC) of plasma neurofilament light in predicting clinical diagnosis | Baseline, 1 year, 2 years, 3 years, 4 years, 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Randall Bateman, MD, Principal Investigator — Washington University School of Medicine; David Carr, MD, Study Director — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified blood biomarker, clinical cognitive assessment, PET, and demographic data will be made available for sharing in the LONI IDA repository. Genetic data (genome-wide associated studies) will be made available in the dbGaP repository.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Shared data generated from this project will be made available as soon as possible, and no later than the time of publication or the end of the funding period, whichever comes first. The duration of preservation and sharing of the data is subject to policies followed by dbGaP and LONI IDA repositories.
Access Criteria: Given the sensitive nature of the dataset, data will be made available in LONI IDA and dbGaP data repositories, which restrict access to the data to qualified investigators with an approved data use agreement (DUA). Data can be accessed after application and approval through the LONI IDA and dbGaP databases.

REFERENCES:
- [Background] Li M, Li Y, Schindler SE, Yen D, Sutcliffe S, Babulal GM, Benzinger TLS, Lenze EJ, Bateman RJ. Design and feasibility of an Alzheimer's disease blood test study in a diverse community-based population. Alzheimers Dement. 2023 Dec;19(12):5387-5398. doi: 10.1002/alz.13125. Epub 2023 May 19. PMID 37204806
- [Background] Janelidze S, Bali D, Ashton NJ, Barthelemy NR, Vanbrabant J, Stoops E, Vanmechelen E, He Y, Dolado AO, Triana-Baltzer G, Pontecorvo MJ, Zetterberg H, Kolb H, Vandijck M, Blennow K, Bateman RJ, Hansson O. Head-to-head comparison of 10 plasma phospho-tau assays in prodromal Alzheimer's disease. Brain. 2023 Apr 19;146(4):1592-1601. doi: 10.1093/brain/awac333. PMID 36087307
- [Background] Janelidze S, Teunissen CE, Zetterberg H, Allue JA, Sarasa L, Eichenlaub U, Bittner T, Ovod V, Verberk IMW, Toba K, Nakamura A, Bateman RJ, Blennow K, Hansson O. Head-to-Head Comparison of 8 Plasma Amyloid-beta 42/40 Assays in Alzheimer Disease. JAMA Neurol. 2021 Nov 1;78(11):1375-1382. doi: 10.1001/jamaneurol.2021.3180. PMID 34542571